CLINICAL TRIAL: NCT04913688
Title: The Learning Curve of Emergency Physicians Performed Point-of-care Lower-extremity Ultrasonography in the Diagnosis of Deep Venous Thrombosis
Brief Title: The Learning Curve of Emergency Physicians Performed Lower-extremity Ultrasonography in the Diagnosis of DVT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-01-128
Record Dates: First submitted 2021-05-30; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- suspected DVT group: If deep vein thrombosis (DVT) is suspected among patients who visit the emergency department, the patients become eligible for study subjects.
  Interventions: Procedure: bedside ultrasound performed group

INTERVENTIONS:
Procedure: bedside ultrasound performed group — If deep vein thrombosis (DVT) is suspected among patients who visit the emergency department, an emergency physician performs bedside ultrasound of lower extremities to the patients agreed to participate in this study. The patients also are examined duplex ultrasound by radiologist.

SUMMARY:
If deep vein thrombosis (DVT) is suspected among patients who have symptoms such as pain or swelling of the lower extremities, duplex ultrasound of the lower limb is the first-line imaging modality to diagnose DVT. However, duplex ultrasound is time consuming, requires patient transport to a diagnostic imaging facility.

In recent years, abbereviated bedside ultrasound technique has been accepted by emergency physician to diagnose the presence of DVT. Several studies have proven that the accuracy of this abbreviated bedsude ultrasound for assessing the presence of deep vein thrombosis is not inferior to experts, but how much ultrasound experience is required to obtain the accuracy that does not inferior to experts has yet to be studied.

The aim of this study is to identify how much learning by emergency physicians is needed to obtain the accuracy of the lower extremity ultrasound examination comparable to that of experts.

DETAILED DESCRIPTION:
If deep vein thrombosis (DVT) is suspected among patients who have symptoms such as pain or swelling of the lower extremities, duplex ultrasound of the lower limb is the first-line imaging modality to diagnose DVT. However, duplex ultrasound is time consuming, requires patient transport to a diagnostic imaging facility, and the immediate availability of a trained radiologist or other vascular physician to provide a result since most physicians are unable to interpret such imaging.

In recent years, abbereviated bedside ultrasound technique has been accepted by emergency physician to diagnose the presence of DVT. Compression is applied to assess the presence of thrombus and collapsibility only in three regions - iliofemoral junction, superficial femoral vein, popliteal vein.

Several studies have proven that the accuracy of this abbreviated bedsude ultrasound for assessing the presence of deep vein thrombosis is not inferior to experts, but how much ultrasound experience is required to obtain the accuracy that does not inferior to experts has yet to be studied.

The aim of this study is to identify how much learning by emergency physicians is needed to obtain the accuracy of the lower extremity ultrasound examination comparable to that of experts.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* Among patients who visited the emergency department with symptoms related to lower extremities (e.g. lower extremity pain, swelling of the lower extremities, numbness of the lower extremities, redness of the lower extremities), the clinician judges that an ultrasonography of the lower extremity is necessary based on the medical history, physical examination, and blood test results.
* (or) Patients who need additional ultrasound of the lower extremity vein to check for deep vein thrombosis due to the detection of a pulmonary thromboembolism in an emergency department

Exclusion Criteria:

* Do not agree to participate in the study
* Patients who refuse ultrasound of the lower extremities by an emergency physician or radiologist
* Patients who have already performed an ultrasound of the lower extremities at another hospital and have been diagnosed with DVT
* Patients with a history of chronic deep vein thrombosis
* Patients with hemodynamic instability to refer to diagnostic imaging facility for duplex exam

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: who visiting an emergency department of tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
The number of ultrasound exams | through study completion, an average of 1 year
  The number of ultrasound exams required until the bedside ultrasound of the lower extremities performed by an emergency physician has adequate proficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Yoon, Professor, Study Chair — Samsung medical center, Emergency department
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No